CLINICAL TRIAL: NCT02763774
Title: Effects of Exercise Rehabilitation Program at Hospitalar Fase on Inflammatory Markers, Functional Capacity and Clinical Outcomes in Patients With Left Ventricular Dysfunction After Coronary Artery Bypass Grafting
Brief Title: Effects a Rehabilitation Program in Patients With Left Ventricular Dysfunction After Coronary Artery Bypass Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Solange Guizilini, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31295914.0.0000.5505
Record Dates: First submitted 2016-04-13; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Disorder; Heart, Functional, Postoperative, Cardiac Surgery
Keywords: coronary artery bypass; sistemic inflammatory response syndrome; left ventricular dysfunction; postoperative complications; physical fitness
MeSH Terms: conditions — Ventricular Dysfunction, Left; Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Walking exercise (Experimental): Participants will be sumitted to progressive exercises and supervised by a physiotherapist, active-assisted to free active exercise in upper and lower limbs, stationary running and walking. The intensity of walk will be determined by the Borg's sujective effort perception scale - (modified from zero to 10). On first postoperative day, participants will perform exercises in supine position. From the second to the fifth postoperative day, they will perform progressive walking.
  Interventions: Other: Walking exercise
- Stationary cycling exercise (Experimental): Participants will be sumitted to progressive exercises and supervised by a physiotherapist, active-assisted to free active exercise in upper and lower limbs. From the first to the fifth postoperative day, they will perform progressive cycling exercise.The intensity of cycling will be determined by the Borg's sujective effort perception scale - (modified from zero to 10).
  Interventions: Other: Stationary cycling exercise
- Neuromuscular electrical stimulation (Experimental): Participants will be sumitted to progressive exercises and supervised by a physiotherapist, active-assisted to free active exercise in upper and lower limbs. From the first to the fifth postoperative day, quadriceps and gastrocnemius muscles will be percutaneous stimulated with the following parameters: Synchronic mode, 50Hz, 400uS, time on 10s, time off 20s, intensity as tolerated by the patient.
  Interventions: Other: Neuromuscular electrical stimulation

INTERVENTIONS:
Other: Walking exercise — Participants will be sumitted to progressive exercises and supervised by a physiotherapist, active-assisted to free active exercise in upper and lower limbs, stationary running and walking. The intensity of walk will be determined by the Borg's sujective effort perception scale - (modified from zero to 10). On first postoperative day, participants will perform exercises in supine position. From the second to the fifth postoperative day, they will perform progressive walking.
  Arms: Walking exercise
Other: Stationary cycling exercise — Participants will be sumitted to progressive exercises and supervised by a physiotherapist, active-assisted to free active exercise in upper and lower limbs. From the first to the fifth postoperative day, they will perform progressive cycling exercise.The intensity of cycling will be determined by the Borg's sujective effort perception scale - (modified from zero to 10).
  Arms: Stationary cycling exercise
Other: Neuromuscular electrical stimulation — Participants will be sumitted to progressive exercises and supervised by a physiotherapist, active-assisted to free active exercise in upper and lower limbs. From the first to the fifth postoperative day, quadriceps and gastrocnemius muscles will be percutaneous stimulated with the following parameters: Synchronic mode, 50Hz, 400uS, time on 10s, time off 20s, intensity as tolerated by the patient.
  Arms: Neuromuscular electrical stimulation

SUMMARY:
This study aims to analyze effects of three types of cardiac rehabilitation protocol on fuctional capacity, inflammatory markers, pulmonary function and clinical outcomes after coronary artery bypass grafting (CABG) in patients with left ventricular disfunction. Patients will be randomized and allocated in three groups according to type of exercise protocol: 1. walk; 2. cycle; 3. functional electrical stimulation.

DETAILED DESCRIPTION:
Several studies have been demonstrated beneficial effects of exercise to minimize impact of CABG. However, there is no consensus on what kind of exercise is safe and effective for patients with left ventricular dysfunction.

Walking

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease proven by coronary angiography;
* Elective CABG;
* No acute or chronic pulmonary disease;
* Patients after surgery, keep in spontaneous ventilation on first postoperative day;
* Absence of neurological, neuromuscular, musculoskeletal and osteoarticular incapacitating;
* Consent form signed for participation in the survey.

Exclusion Criteria:

* Inability to perform spirometry;
* Presence of acute lung disease or chronic;
* Surgical indication of urgency;
* Morbid obesity;
* Hemodynamics instability at the time of spirometry or during six minutes walking test;
* Intraoperative death or until the sixth postoperative day;
* Patients remaining in mechanical prolonged ventilation for more than 12 hours;
* Severe cardiac arrhythmia during application of assessment protocols and exercises (ventricular tachycardia, atrioventricular block second or degree) any other condition the investigator's discretion put the patient at increased risk with beginning of the year; Any change that may lead to failure of proposed protocols.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | Up to ten days after surgery, at hospital discharge.
  Participants will be submitted to six minute walk test on preoperative period and sixth postoperative day (or before hospital discharge) to evaluate functional capacity. The test will be performed with a mobile device to measure metabolic response to exercise (Oxycon™ Mobile).

SECONDARY OUTCOMES:
Inflammatory markers | in-hospital postoperative period, up to ten days after surgery.
  Blood sample will be collected to measure inflammatory markers (TNF-alpha and interleukins) and to compare exercise effects on inflammatory response after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Solange Guizilini, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes